CLINICAL TRIAL: NCT04605107
Title: Comparative Randomized, Single Dose, Parallel, Triple-blinded Study in Infertile Females to Evaluate Biosimilarity of IM Injection of Human Chorionic Gonadotrophin After Parenteral Administration of Treatment A TEST Product Epifasi 5000 I.U. Ampoules (EIPICO PHARMA, EGYPT) and Treatment B REFERENCE Product Pregnyl 5000 I.U. Ampoules (Baxter Pharmaceutical Solutions for Organon, USA)
Brief Title: Biosimilarity Study of IM Injection of Human Chorionic Gonadotrophin After Parenteral Administration of Treatment A TEST Product Epifasi 5000 I.U. Ampoules (EIPICO PHARMA, EGYPT) and Treatment B REFERENCE Product Pregnyl 5000 I.U. Ampoules (Baxter Pharmaceutical Solutions for Organon, USA).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: EIPICO PHARMA, EGYPT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GRC/1/13/433
Record Dates: First submitted 2020-09-22; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-09

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A test (Experimental): Epifasi 5000 I.U. Ampoules
  Interventions: Drug: Epifasi: Human chorionic gonadotrophin
- B reference (Active Comparator): Pregnyl 5000 I.U. Ampoules
  Interventions: Drug: Pregnyl: Human chorionic gonadotrophin

INTERVENTIONS:
Drug: Epifasi: Human chorionic gonadotrophin — IM Injection of 1 ampoule contains 5000 I.U. of Human chorionic gonadotrophin
  Other Names: Epifasi
  Arms: A test
Drug: Pregnyl: Human chorionic gonadotrophin — IM Injection of 1 ampoule contains 5000 I.U. of Human chorionic gonadotrophin
  Other Names: Pregnyl
  Arms: B reference

SUMMARY:
Comparative randomized, single dose, parallel, triple-blinded study in infertile females to evaluate biosimilarity of IM Injection of Human Chorionic Gonadotrophin (HCG) after Parenteral administration of Treatment A TEST Product Epifasi 5000 I.U. Ampoules (EIPICO PHARMA, EGYPT) and Treatment B REFERENCE Product Pregnyl 5000 I.U. Ampoules (Baxter Pharmaceutical Solutions for Organon, USA)

DETAILED DESCRIPTION:
In this study, the biosimilarity of Human chorionic gonadotropin (HCG) from Epifasi IM Injection (EIPICO Pharma Egypt) and Pregnyl IM Injection (Baxter Pharmaceutical Solutions for Organon, USA) after a single IM dose administration of each to healthy adult will be investigated to determining the study variables: Ovarian Ultrasonic counting mature grafian follicles, Number of retrieved oocytes and their grades.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal woman between 18 - 40 years of age.
2. Body mass index (BMI) of 32 or less.
3. A menstrual cycle lasting between 21 and 35 days.
4. Serum hormone levels of FSH 12 IU/L or less, PRL 1040 mIU/L or less, and TSH within the normal range of 0.3- 4.9 mIU/L
5. Patient having both ovaries and a normal uterine cavity confirmed by hysteroscopy, or hysterosalpingography.
6. All patients had to be infertile due to at least one of the following causes and must have justified ART (Assisted Reproductive Technology) treatment: tubal factor, mild endometriosis (American Fertility Society classification stage I orII), unexplained infertility, or male factor
7. Patients achieving good ovarian response and considered to receive hCG for final follicular maturation prior to OPU.
8. Written and signed informed consent by the patient.
9. Subject does not have allergy to the drugs under investigation.
10. Medical demographics without evidence of clinically significant deviation from rather normal medical condition.

Exclusion Criteria:

1. Patients with low ovarian reserve, as proved by hormonal assays and basal antral follicular count.
2. More than three previous assisted reproductive technology cycle or treatment with clomiphene citrate or gonadotropins for at least 1 month before screening,
3. Patients with pelvic abnormality that would interfere with ovarian accessibility for OPU, e.g. ovarian endometriotic cysts or high and retro-uterine ovary.
4. Patients not achieving a satisfactory ovarian response on ovulation induction, whether poor response (3 or less mature ovarian follicles) or over-response with high likelihood of developing ovarian hyperstimulation syndrome (OHSS) on triggering with HCG.
5. History of hypersensitivity to the study medications or to drugs with similar chemical structure.
6. Patients unlikely to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and likelihood of not completing the study.
7. Mental condition rendering the patients unable to understand the nature, scope and possible consequences of the study.
8. Results of laboratory tests which are clinically significant.
9. Acute infection within one week preceding first study drug administration.
10. History of drug or alcohol abuse.
11. Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
12. Subject is on a special diet (for example subject is vegetarian).
13. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
14. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
15. Subject has a history of severe diseases which have direct impact on the study.
16. Participation in a biosimilarity study or in a clinical study within the last 6 weeks before first study drug administration.
17. Subject intends to be hospitalized within 3 months after first study drug administration.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile and anovulatory females of age 18-40 years, BMI ≤32, Menstrual cycle lasting between 21-35 days, Hormones (FSH, PRL and TSH) within normal levels, two ovaries and a normal uterine cavity and Justified for ART as a result of tubal factor, mild endometriosis, unexplained or male factor.
Enrollment: 60 (Actual)
Dates: Start 2013-08-30 (Actual); Primary Completion 2015-01-08 (Actual); Study Completion 2015-03-08 (Actual)

PRIMARY OUTCOMES:
No. of mature follicles | Up to 34-36 hours post dose
  A dose of Epifasi 5000 I.U. Ampoule was injected to trigger ovulation., At least, one mature follicle should be detected with a diameter of 18 mm or more & two additional follicles reached a diameter of 16 mm or more. 34 to 36 hours later oocytes were retrieved.

SECONDARY OUTCOMES:
Safety Evaluation | the patient is observed during the whole course of the study and for one month post study
  Any reported adverse effect from the patient side or observed by the investigator, Also any abnormal lab finding.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — Genuine Research Center
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steinijans VW, Diletti E. Statistical analysis of bioavailability studies: parametric and nonparametric confidence intervals. Eur J Clin Pharmacol. 1983;24(1):127-36. doi: 10.1007/BF00613939. PMID 6832195
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Background] Driscoll GL, Tyler JP, Hangan JT, Fisher PR, Birdsall MA, Knight DC. A prospective, randomized, controlled, double-blind, double-dummy comparison of recombinant and urinary HCG for inducing oocyte maturation and follicular luteinization in ovarian stimulation. Hum Reprod. 2000 Jun;15(6):1305-10. doi: 10.1093/humrep/15.6.1305. PMID 10831560
- See also: International conference of harmonization of technical requirements for registration of pharmaceuticals for human use. ICH harmonized tripartite guideline. Guidelines for good clinical practice. May 1996. — http://www.pharmaweb.net/pwmirror/pw9/ifpma/ich1.html
- See also: The European Agency for the Evaluation of Medicinal products (EMEA). Note for guidance on good clinical practice (CPMP/ICH/135/95), May 1997. — https://www.ema.europa.eu
- See also: Guidance for Industry: Bioavailability and Bioequivalence studies for orally administered drug products-general considerations. US Dept. of Health and Human Services, food and drug administration (FDA), center for drug evaluation and research (CDER), M — https://www.fda.gov/drugs/guidance-compliance-regulatory-information